CLINICAL TRIAL: NCT02030626
Title: Comparison of the Efficacy of Repetitive Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation of the Motor Cortex in Patients With Neuropathic Pain Due to Chronic Radiculopathy
Brief Title: Comparison of the Efficacy of rTMS and tDCS of the Motor Cortex in Patients With Chronic Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, MD PhD, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTMS versus tDCS; 2010-018309-12 (Registry Identifier: eudract)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Lumbar Radiculopathy
Keywords: Neuropathic pain; lumbar radiculopathy; rTMS; tDCS; placebo controlled study
MeSH Terms: conditions — Radiculopathy; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active rTMS or active tDCS or placebo (Experimental): Active rTMS (10 Hz) of the motor cortex followed by active tDCS (2 mA) of the motor cortex or conversely
  Interventions: Device: active or placebo rTMS or active or placebo tDCS
- Sham rTMS followed by tDCS (or conversely) (Placebo Comparator): Placebo rTMD followed by placebo tDCS or conversely
  Interventions: Device: active or placebo rTMS or active or placebo tDCS

INTERVENTIONS:
Device: active or placebo rTMS or active or placebo tDCS

SUMMARY:
The present study aims to compare directly the efficacy of two noninvasive neurostimulation techniques : repetitive transcranial magnetic stimulation and transcranial direct electrical current of the motor cortex in patients with chronic lumbar radiculopathy on pain intensity.

DETAILED DESCRIPTION:
The present study ims to compare directly the efficacy of two noninvasive neurostimulation techniques : repetitive transcranial magnetic stimulation (rTMS) and transcranial direct electrical current (tDCS) of the motor cortex in patients with chronic lumbar radiculopathy on average pain intensity. This will be a sham controlled crossover design : patients will be randomized to receive either active rTMS or tDCS during 3 consecutive days followed by the alternative treatment within 3 weeks apart, or sham rTMS or tDCS during 3 consecutive dats followed by the alternative treatment within 3 weeks apart. The investigator will be blind to the treatment. Assessments will be performed before each treatment, then 1 hour after the end of the third day session, then 2 days and 1 week after the stimulation. Assessments will include pain questionnaires, quality of life, anxiety and depression, catastrophizing and evaluation of treatment effect on experimental pain using Quantitative sensory testing.

ELIGIBILITY:
Inclusion Criteria:

Patients aged more than 18 years and less than 60 years, males of females Lumbosciatica or lumbocruralgia with predominant neuropathic components with DN4 score ≥ 4/10 Chronic pain with an intensity of at least 4/10 Stable analgesic treatment for at least 15 days before inclusion Able to speak and understand French Social security

Exclusion Criteria:

Work accident or litigation Contraindication to rTMS (sismotherapy in the preceding month, epilepsia, past head trauma, intracranial hypertension, metallic clip, pace maker, pregnancy or lactation Major depressive episode Intermittent pain Consent refusal Impossible to follow up during the duration of the study Pain more severe than neuropathic pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Comparison of rTMS and tDCS on average pain intensity | 7 days after 3 days of stimulation
  Average pain intensity numerical scales (0-10)

SECONDARY OUTCOMES:
Comparison of rTMS and sham stimulation on average pain intensity | 7 days after 3 stimulation days
  numerical scale for pain intensity (0-10)
comparison of tDCS and sham stimulation on average pain intensity | at 7 days after 3 days of stimulation
  numerical scales for pain intensity (0-10)
comparison of rTMS and tDCS on current pain | 1 hour after each stimulation session
  pain intensity (right now)1 hour after each stimulation
comparison of rTMS and tDCS on pain intensity | 2 days after 3 stimulation days
  numerical score (0-10) for pain over the last 24 hours
comparison of rTMS versus tDCS and versus sham on BPI interference | 7 days after the end of 3 stimulation days
  BPI interference scale (0-70)
comparison of rTMS versus tDCS and sham on pain catastrophizing | 7 days after the last day of stimulation (3 days)
  Pain catastrophizing scale (PCS)
comparison of rTMS versus tDCS and sham on anxiety and depression | 7 days after the end of stimulation sessions
  Hospital anxiety and depression scale
comparison of rTMS versus tDCS and sham on neuropathic symptoms | 7 days after the end of stimulations
  Neuropathic pain symptom inventory
comparison of rTMS versus tDCS and sham on thermal testing | 2 days and 7 days after stimulation days
  thermal testing using thermotest on the upper limbs
comparison of safety between rTMS and tDCS and between neurostimulation and sham | immediately after each stimulation, then at 2 days and 7 days
  any emerging side effects

CONTACTS AND LOCATIONS:
Overall Officials: Didier BOUHASSIRA, MD PhD, Study Director — INSERM U 987; Jean Pascal LEFAUCHEUR, MD PhD, Principal Investigator — APHP
Locations (2):
- France (2):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Henri Mondor, APHP, Créteil